CLINICAL TRIAL: NCT03352726
Title: An Open-label Phase I Study to Assess the Biological Potency of Peanut Allergen Extract in Adolescent and Adult Peanut Allergic Subjects
Brief Title: A Study to Assess the Biological Potency of Peanut Allergen Extract in Adolescent and Adult Peanut Allergic Subjects
Acronym: V712-103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIOPOT
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Peanut Allergy
Keywords: EPIT; Epicutaneous; Immunotherapy; Viaskin
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DBV712 Solution for Skin Prick Test (Experimental): DBV712 In-House Reference Skin Prick Test preparation
  Interventions: Drug: DBV712 IHRP

INTERVENTIONS:
Drug: DBV712 IHRP — DBV712 Solution for Skin Prick Test

SUMMARY:
The study aims to assess the biological potency of the In-House Reference Preparation (IHRP) of peanut allergens extract by a quantitative Skin Prick Test (SPT) method in peanut-allergic subjects.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female subjects aged between 12-50 years
* Physician-diagnosed peanut allergy
* Subject currently following a strict peanut-free diet
* Documented history of positive test to peanut-specific IgE (ImmunoCAP system) >0.7 kU/L
* Positive peanut SPT with a largest wheal diameter ≥ 8 mm

Main Exclusion Criteria:

* Uncontrolled asthma
* Peanut allergen immunotherapy whatever the route, either ongoing or previously started and having lasted more than one month (>30 days)
* Topical use of steroids within the past 14 days prior to the Screening SPT
* Inability to discontinue short-acting antihistamines
* Atopic dermatitis, eczema or urticaria on the areas to be tested

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Biological potency of the In-House Reference peanut proteins extract (DBV712-IHRP) in arbitrary Biological Units (BU) | 1 day to 2 weeks

SECONDARY OUTCOMES:
Adverse Events (AEs), Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) | Throughout the study (1 day to 2 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado